CLINICAL TRIAL: NCT06617936
Title: Tislelizumab Combined With Recombinant Human Endostatin Injection Plus Chemotherapy in Unresectable Stage III NSCLC: a Prospective, Single-arm, Multicenter Phase II Clinical Study
Brief Title: Tislelizumab Combined With Recombinant Human Endostatin Combined With Chemotherapy for Unresectable Stage III Non-small Cell Lung Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hua Zhang (Other Government)
Responsible Party: Sponsor-Investigator, Hua Zhang, Head of thoracic surgery, Shandong Public Health Clinical Center
Organization: Shandong Public Health Clinical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GWLCZXEC2024-55-2
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Unresectable Non-small Cell Lung Cancer
Keywords: neoadjuvant therapy; NSCLC; immunotherapy
MeSH Terms: interventions — Drug Therapy; Surgical Procedures, Operative; Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant Group/Arm A (Experimental): Participants receive 2-4 cycles of Tislelizumab With Recombinant human endostatin combined with Chemotherapy treatment during preoperative period, every 3 weeks once for 4 cycles at most.
  After neoadjuvant therapy, Patients evaluated for MDT who can be surgically resected will be placed in the surgical group for surgical excision.
  Surgery will be performed within 4 to 6 weeks after completion of preoperative therapy.
  After surgery, participants will receive adjuvant therapy with tislelizumab combined with recombinant human endostatin injection every 3 weeks until disease progression or postoperative adjuvant therapy for 1 year.
  Interventions: Drug: neoadjuvant therapy:Tislelizumab With Recombinant human endostatin combined with Chemotherapy; Procedure: surgery; Drug: Adjuvant therapy:Tislelizumab and Recombinant Human Endostatin Injection (Endostar)
- Participant Group/Arm B (Experimental): Participants receive 2-4 cycles of Tislelizumab With Recombinant human endostatin combined with Chemotherapy treatment , every 3 weeks once for 4 cycles at most. After neoadjuvant therapy, Patients evaluated by MDT as unresectable will be placed in the standard treatment group, where the investigator will select the standard treatment regimen determined by the MDT discussion.
  Interventions: Drug: neoadjuvant therapy:Tislelizumab With Recombinant human endostatin combined with Chemotherapy; Other: Standard Treatment

INTERVENTIONS:
Drug: neoadjuvant therapy:Tislelizumab With Recombinant human endostatin combined with Chemotherapy — neoadjuvant therapy : Tislelizumab: 200mg, ivgtt, day 1 ; Recombinant Human Endostatin Injection (Endostar),210mg was pumped intravenously for 3 consecutive days; Pemetrexed (Non-squamous NSCLC) or Nab-paclitaxel(Squamous NSCLC):Pemetrexed: 500 mg/m^2, ivgtt, day 1. Nab-paclitaxel: 260mg/m^2, ivgtt, day 1.; Carboplatin:Carboplatin was given dosed to an area under the serum concentration-time curve (AUC) of 5 ivgtt on day 1 ; every 21 days for 1 cycle,2-4 cycles; (If the preoperative neoadjuvant did not reach 4 cycles, the treatment with ralizumab combined with recombinant human endostatin injection and chemotherapy for 1-2 cycles can be continued after surgery, and the total cycle of chemotherapy before and after surgery is up to 4 cycles)
Procedure: surgery — Patients who are discussed by the MDT panel to evaluate surgical resection will undergo surgery.Surgery must be done within the 4th-6th week from day 1 the last cycle of neoadjuvant treatment.
  Arms: Participant Group/Arm A
Drug: Adjuvant therapy:Tislelizumab and Recombinant Human Endostatin Injection (Endostar) — Adjuvant therapy Tislelizumab: 200mg, ivgtt, day 1 of each 21-day cycle, 17 cycles at most. Recombinant Human Endostatin Injection (Endostar):210mg was pumped intravenously for 3 consecutive days, every 21 days for 1 cycle,17 cycles at most.
  Arms: Participant Group/Arm A
Other: Standard Treatment — Patients assessed by the MDT panel as inoperable for surgical treatment will be selected by the investigator for a standard treatment protocol determined by the MDT discussion
  Arms: Participant Group/Arm B

SUMMARY:
This is a prospective, single-arm, multicenter, phase II clinical study designed to evaluate the initial efficacy and safety of patients receiving Tislelizumab in combination with recombinant human endostatin injection plus chemotherapy for stage III unresectable non-small cell lung cancer. To evaluate the surgical conversion rate of tirellizumab combined with recombinant human endostatin injection and chemotherapy induction therapy in patients with initially unresectable stage III non-small cell lung cancer.

ELIGIBILITY:
1. Have fully understood the study and voluntarily signed the informed consent;
2. Age 18-75 years old, gender is not limited;
3. Histologically confirmed Stage III initial unresectable squamous or non-squamous non-small cell lung cancer (AJCC Stage 8th edition)

   - Unresectable stage III NSCLC mainly refers to imaging or lymph node pathological evidence: Multiple metastases of ipsilateral mediastinal lymph nodes fused into masses or multisite metastases (IIIA: T1-2N2 or IIIB: T3-4N2); metastases to the contralateral hilar, mediastinal lymph nodes, or to the same, contralateral scalene, or supraclavicular lymph nodes (IIIB: T1-2N3, IIIC: T3-4N3); lesion invasion of important organs (including diaphragm, mediastinum, great blood vessels, trachea, recurrent laryngeal nerve, esophagus, or satellite nodules in different pulmonary lobes on the same side of the primary tumor, resulting in clinician determination that R0 resection could not be performed) (IIIA: T4N0-1); Determination of o N2/N3 lymph node involvement: PET-CT was used to confirm lymph node status. In cases where PET-CT is insufficient to determine lymph node staging (for example, lymph node diameter <2cm), pathologic confirmation (EBUS/EUS/ thoracoscopic/mediastinoscopy or fine needle aspiration biopsy) is performed by the investigator to select appropriate lymph nodes to determine the staging.

   Clinical evaluation of unresectable Stage III NSCLC: Other clinicians determine that R0 resection is not feasible or that a total lung resection is required to achieve R0 resection.
4. At least 1 measurable lesion as defined by RECIST v1.1;
5. ECOG score 0-1;
6. Eligible for platinum-containing double-drug chemotherapy.
7. Good organ function;

   • Patients have not received blood transfusion or growth factor support therapy ≤ 14 days prior to sample collection during the screening period and: Absolute neutral cell count (ANC) ≥1.5 x 109/L
   * Platelet ≥100 x 109/L
   * Hemoglobin ≥90 g/L

     • Calculated creatinine clearance (CrCl) (Cockcroft-Gault formula)
   * Patients scheduled to receive cisplatin: creatinine clearance ≥ 60 mL/min
   * Patients scheduled to receive carboplatin: creatinine clearance ≥ 45 mL/min

     * Serum total bilirubin ≤1.5 × upper limit of normal (ULN) (patients with Gilbert's syndrome must have total bilirubin < 3 × ULN)
     * AST and ALT≤ 2.5 x ULN
     * Patients who did not receive anticoagulant therapy: International standardized ratio or activated partial thromboplastin time ≤ 1.5 × ULN
     * Albumin ≥25 g/L (2.5 g/dL).
8. Willing and able to comply with study plan visits, treatment plans, laboratory tests and other study procedures;
9. The total amount of lung function, as assessed by the surgeon, is sufficient to withstand the proposed pneumonectomy;
10. Women of childbearing age must take a serum pregnancy test within 3 days before the first medication, and the result is negative. Female subjects of reproductive age and male subjects whose partners are women of reproductive age must agree to use highly effective methods of contraception during the study period and for 120 days after the last dose of the study drug

Exclusion Criteria:

1. Patients with known EGFR gene mutation, ALK rearrangement, ROS-1 fusion, RET fusion, HER-2 mutation, MET mutation, and non-squamous cell carcinoma with unknown driver gene status;
2. Previous treatment for current lung cancer, including radiotherapy and all systemic antitumor agents, including chemotherapy, immunotherapy, targeted therapy or antiangiogenic therapy.
3. Patients with large cell neuroendocrine carcinoma (LCNEC) components and non-small cell lung cancer with mixed small cell components.
4. Patients received other approved systemic immunomodulators (including, but not limited to, interferon, interleukin 2, tumor necrosis factor, thymus pentapeptide, and thymofasin) within 4 weeks prior to initial administration.
5. In the course of treatment, researchers determined that patients' tumors were more likely to invade important blood vessels and cause fatal bleeding.
6. Clinically significant hemoptysis (more than 50ml of hemoptysis per day), or clinically significant bleeding symptoms or significant bleeding tendency (such as gastrointestinal bleeding, gastric ulcer bleeding, gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occulted blood ++ or above baseline, or vasculitis) within 3 months before the study.
7. Any Chinese herbs used for cancer control were used within 14 days prior to the first administration of the study drug.
8. Have received live vaccine within 30 days before the first dose. Including but not limited to the following: mumps, rubella, measles, varicella/shingles (chickenpox), yellow fever, rabies, BCG and typhoid vaccine (inactivated virus vaccine allowed); Live or attenuated vaccine is expected to be required during the study period or within 5 months after the last dose.
9. For any condition requiring systemic treatment with corticosteroids (prednisone or equivalent >10 mg/ day) or other immunosuppressive agents within 14 days prior to the first administration of the study drug, the investigator assessed the patient as having an impact on the study treatment.
10. Active autoimmune diseases requiring systemic treatment in patients assessed by the investigator as having an impact on investigational treatment.
11. Patients with interstitial lung disease, non-infectious pneumonia, or other diseases that are not under control, including diabetes, pulmonary fibrosis, acute lung disease, etc., that the investigators have assessed as having an impact on the study treatment.
12. Patients with a history of major diseases or clinical manifestations that may affect the function of organ systems and are assessed by the investigator as having implications for the study and treatment.
13. Study severe chronic or active infections (including tuberculosis) requiring systemic antimicrobial, antifungal, or antiviral treatment ≤14 days before the first administration of the drug.
14. Uncontrolled active hepatitis B (defined as positive HBV surface antigen [HBsAg] test results during screening and HBV-DNA test values higher than the upper limit of normal values in the laboratory of the research center; (Participants with HBV-DNA levels < 500 IU/mL within 28 days prior to enrollment, who have received local standard antiviral therapy for at least 14 days and who are willing to continue antiviral therapy during the study period may be enrolled); Subjects with active hepatitis C (defined as positive HCV surface antibody [HCsAb] test results during screening, positive HCV-RNA);
15. Known human immunodeficiency virus (HIV) infection (known HIV antibody positive);
16. Grade III-IV congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmias;
17. Any arterial thrombosis, embolism, or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, occurred within 6 months prior to treatment;
18. Concurrent participation in another therapeutic clinical study, unless it is an observational (non-interventional) clinical study or in the follow-up period of an interventional study.
19. Medical history or evidence of disease that may interfere with the test results, prevent participants from participating fully in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment. The Investigator considers that there are other potential risks that are not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Surgical resection rate | From enrollment to the end of surgery
  Proportion of patients who underwent surgical resection after induction therapy

SECONDARY OUTCOMES:
Objective response rate (ORR) | prior to surgery
  ORR is defined as the percentage of participants having a complete response or a partial response, measured by RECIST 1.1.
Event-Free Survival(EFS) | Up to 2years
  The time from the start of randomization (or the start of treatment in a one-arm trial) to the first occurrence of any of the following events: disease progression without surgical treatment, local or distant recurrence, death from any cause, etc.
Pathological Complete Response (pCR) Rate | 1 month after surgery
  no residual tumor cells in the surgically resected tumor specimen and all sampled regional lymph nodes after neoadjuvant treatment.
Major Pathological Response (MPR) Rate | 1 month after surgery
  Major Pathological Response (MPR) Rate: defined as ≤ 10% of residual tumor cells in the surgically resected tumor specimen and sampled regional lymph nodes after neoadjuvant treatment.
Progression-Free Survival (PFS) | Up to 12 months
  Progression-Free Survival (PFS): defined as the time from the first dose until the date of first documented progression or date of death from any cause, whichever came first.
Overall Survival | 3 years
  Time from randomization to death (from any cause)
1 years event free survival (EFS) | 1 years
  1 years EFS rate is defined as the percentage of participants having no radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause within 1years after randomization.
1 years Progression-Free Survival (PFS) | 1 years after randomization
  1 years Progression-Free Survival (PFS): defined as the time from the first dose until the date of first documented progression or date of death from any cause, whichever came first within 1 years after randomization.
1 years overall survival rate (OS) | 1 years after randomization
  1 years OS rate is defined as the percentage of participants having no death of any cause within 1 years after operation.The Kaplan-Meier estimator will be used to estimate median OS and its 95%CI and the survival curve.
R0 Resection Rate | 1 month after surgery
  R0 Resection Rate: The pathological results will showed that the incision margin was negative and no residual cancer cells were found under the microscope.
Safety and Tolerability | Up to 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Public Health Clinical Center (ShandongPHCC), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Protect patient privacy